CLINICAL TRIAL: NCT00877890
Title: A Randomized, Open-Label, Parallel-Group, Comparator-Controlled, Multicenter Study to Evaluate the Glycemic Effects, Safety, and Tolerability of Exenatide Once Weekly in Subjects With Type 2 Diabetes Mellitus
Brief Title: A Study to Evaluate the Glycemic Effects, Safety, and Tolerability of Exenatide Once Weekly in Subjects With Type 2 Diabetes Mellitus (DURATION-5)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCB108 (DURATION-5)
Record Dates: First submitted 2009-04-06; First posted 2009-04-08 (Estimated); Results first posted 2012-06-19 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; exenatide once weekly; Byetta; Amylin; Lilly; Bydureon
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: exenatide once weekly
- 2 (Active Comparator)
  Interventions: Drug: exenatide twice daily

INTERVENTIONS:
Drug: exenatide once weekly — subcutaneous injection, 2.0mg, once a week
  Other Names: BYDUREON
  Arms: 1
Drug: exenatide twice daily — subcutaneous injection; 5mcg (4 weeks) and 10mcg (20 weeks); twice a day
  Other Names: BYETTA
  Arms: 2

SUMMARY:
This study will compare the effects of commercially manufactured exenatide once weekly and exenatide BID in subjects whose type 2 diabetes is managed with diet and exercise alone or with oral antidiabetic medications. The study will examine glycemic control (as measured by HbA1C), safety, and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Has been diagnosed with type 2 diabetes mellitus
* Has hemoglobin-specific A1c fraction (HbA1c) of 7.1% to 11.0%, inclusive, at screening
* Has a body mass index (BMI) of 25 kg/m2 to 45 kg/m2, inclusive, at screening
* Has been treated with diet and exercise alone or in combination with a stable regimen of metformin (MET), a sulfonylurea (SU), a thiazolidinedione (TZD), a combination of metformin and an SU, a combination of metformin and a TZD, or a combination of an SU and a TZD for a minimum of 2 months prior to screening
* Either is not treated with or has been on a stable treatment regimen with any of the following medications for a minimum of 2 months prior to screening:

  * Hormone replacement therapy (female subjects)
  * Oral contraceptives (female subjects)
  * Antihypertensive agents
  * Lipid-lowering agents
  * Thyroid replacement therapy
  * Antidepressant agents
  * Drugs known to affect body weight, including prescription medications (e.g. orlistat [XENICAL®], sibutramine [MERIDIA®], topiramate [TOPAMAX®]) and over the counter antiobesity agents

Exclusion Criteria:

* Has ever been exposed to exenatide (exenatide once weekly [exenatide LAR], exenatide BID, BYETTA, or any other formulation) or any glucagon-like peptide-1 (GLP-1) analog
* Has received any investigational drug within one month (or five half-lives of the investigational drug, whichever is greater) of screening
* Has been treated, is currently being treated, or is expected to require or undergo treatment with any of the following treatment excluded medications:

  * Any dipeptidyl peptidase 4 (DPP-4) inhibitor within 3 months prior to screening
  * Alpha glucosidase inhibitor, meglitinide, nateglinide, or pramlintide (SYMLIN®) within 30 days of screening
  * Insulin within 2 weeks of screening or for more than 1 week within 3 months of screening
  * Systemic corticosteroids by oral, intravenous, or intramuscular route; or potent, inhaled, or intrapulmonary (including ADVAIR®) steroids known to have a high rate of systemic absorption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2009-03; Primary Completion 2009-10 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Porter, MD, Study Director — Amylin Pharmaceuticals, LLC.
Locations (41):
- United States (41):
  - Research Site, Birmingham, Alabama
  - Research Site, Mesa, Arizona
  - Research Site, Peoria, Arizona
  - Research Site, Artesia, California
  - Research Site, Concord, California
  - Research Site, Encino, California
  - Research Site, Greenbrae, California
  - Research Site, La Mesa, California
  - Research Site, Walnut Creek, California
  - Research Site, DeLand, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Miami, Florida
  - Research Site, New Port Richey, Florida
  - Research Site, Palm Harbor, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Avon, Indiana
  - Research Site, Evansville, Indiana
  - Research Site, Lexington, Kentucky
  - Research Site, Paducah, Kentucky
  - Research Site, Detroit, Michigan
  - Research Site, Edina, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Butte, Montana
  - Research Site, New Hyde Park, New York
  - Research Site, Rochester, New York
  - Research Site, Raleigh, North Carolina
  - Research Site, Statesville, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Delaware, Ohio
  - Research Site, Mentor, Ohio
  - Research Site, Eugene, Oregon
  - Research Site, Rapid City, South Dakota
  - Research Site, Austin, Texas
  - Research Site, Corpus Christi, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Burke, Virginia
  - Research Site, Manassas, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Olympia, Washington
  - Research Site, Spokane, Washington
  - Research Site, Tacoma, Washington

REFERENCES:
- [Result] Blevins T, Pullman J, Malloy J, Yan P, Taylor K, Schulteis C, Trautmann M, Porter L. DURATION-5: exenatide once weekly resulted in greater improvements in glycemic control compared with exenatide twice daily in patients with type 2 diabetes. J Clin Endocrinol Metab. 2011 May;96(5):1301-10. doi: 10.1210/jc.2010-2081. Epub 2011 Feb 9. PMID 21307137
- [Derived] Blevins T, Ruggles J, Hardy E. Onset of Glycemic and Weight Outcomes in Patients Initiating Exenatide Once Weekly: The Relationship of Exenatide Exposure with Efficacy over the First 24 Weeks of Treatment. Diabetes Ther. 2016 Jun;7(2):361-8. doi: 10.1007/s13300-016-0172-0. Epub 2016 May 5. PMID 27146799
- [Derived] Grimm M, Han J, Weaver C, Griffin P, Schulteis CT, Dong H, Malloy J. Efficacy, safety, and tolerability of exenatide once weekly in patients with type 2 diabetes mellitus: an integrated analysis of the DURATION trials. Postgrad Med. 2013 May;125(3):47-57. doi: 10.3810/pgm.2013.05.2660. PMID 23748506
- [Derived] Peyrot M, Bushnell DM, Best JH, Martin ML, Cameron A, Patrick DL. Development and validation of the self-management profile for type 2 diabetes (SMP-T2D). Health Qual Life Outcomes. 2012 Oct 5;10:125. doi: 10.1186/1477-7525-10-125. PMID 23039868
- [Derived] Fineman MS, Mace KF, Diamant M, Darsow T, Cirincione BB, Booker Porter TK, Kinninger LA, Trautmann ME. Clinical relevance of anti-exenatide antibodies: safety, efficacy and cross-reactivity with long-term treatment. Diabetes Obes Metab. 2012 Jun;14(6):546-54. doi: 10.1111/j.1463-1326.2012.01561.x. Epub 2012 Feb 10. PMID 22236356

RESULTS

PARTICIPANT FLOW:
Groups:
- Exenatide Once Weekly: Subcutaneous injection of 2 mg exenatide, once a week
- Exenatide Twice Daily: Subcutaneous injection of exenatide, twice a day (5 mcg exenatide per dose for first 4 weeks, then 10 mcg exenatide per dose for 20 weeks)
Period: Overall Study
Arm/Group | Exenatide Once Weekly | Exenatide Twice Daily
Started | 129 | 125
Intent to Treat (ITT) | 129 | 123
Completed | 109 | 95
Not Completed | 20 | 30
Not completed — Adverse Event | 6 | 6
Not completed — Lost to Follow-up | 5 | 5
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal of Consent | 6 | 12
Not completed — Investigator Decision | 0 | 2
Not completed — Loss of Glucose Control | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exenatide Once Weekly | Exenatide Twice Daily | Total
Number analyzed (Participants) | 129 | 123 | 252
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 103 | 102 | 205
  >=65 years | 26 | 21 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (11.14) | 55.2 (10.27) | 55.7 (10.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 55 | 107
  Male | 77 | 68 | 145
Glycosylated hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of total hemoglobin] | 8.5 (1.10) | 8.4 (1.23) | 8.4 (1.16)
Weight [Mean (Standard Deviation); unit: kg] | 97.0 (20.66) | 94.3 (18.94) | 95.7 (19.85)
Background Oral Antidiabetic Agent [Number; unit: participants]
  Diet and Exercise | 21 | 26 | 47
  Metformin (MET) | 51 | 52 | 103
  Sulfonylurea (SU) | 1 | 8 | 9
  Thiazolidinediones (TZD) | 4 | 2 | 6
  MET+SU | 34 | 25 | 59
  MET+TZD | 13 | 9 | 22
  SU+MET+TZD | 5 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline to Week 24
Description: Change in HbA1c from baseline (Day 1) to Week 24 [Week 24 - Baseline].
Time Frame: Day 1, Week 24
Population: The ITT Population consisted of all randomized subjects who received at least one injection of study medication. Missing data up to Week 24 were imputed using the last observation carried forward (LOCF) approach for subjects who had data for at least one scheduled visit (including Early Termination) subsequent to the baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: percentage of total hemoglobin
Arm/Group | Exenatide Once Weekly | Exenatide Twice Daily
Number analyzed (Participants) | 126 | 116
percentage of total hemoglobin | -1.57 (0.104) [-1.77 to -1.36] | -0.90 (0.110) [-1.12 to -0.69]
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Exenatide Twice Daily; Superiority of exenatide once weekly to BYETTA if the upper limit of the 2-sided 95% CI for treatment difference (exenatide once weekly minus BYETTA) is <0; noninferiority if this upper limit is <0.4%. Power: Assuming 15% dropout rate with 206 subjects will complete the study. This sample size would provide 90% power for non-inferiority test with assumption of greater reduction (0.1%) in exenatide once weekly and a common standard deviation of 1.1%; Test type: Non-Inferiority or Equivalence — The choice of a 0.4% noninferiority margin was resulted from the considerations of expected clinical benefit of BYETTA in this study based on clinical data evaluating exenatide once weekly and BYETTA, regulatory guidance, published literature, and statistical considerations; p < .0001, ANOVA; Analysis of variance (ANOVA) model includes treatment, baseline HbA1c stratum (<9% or >=9%), and concomitant SU use at screening as factors; Least Squares Mean Difference = -0.67, 95% CI 2-sided [-0.94 to -0.39], Standard Error of Mean 0.138

2. Secondary Outcome: Percentage of Subjects Achieving HbA1c Target of <7%
Description: Percentages of subjects achieving HbA1c target value of <7% at Week 24.
Time Frame: Week 24
Population: ITT Population. Missing data up to Week 24 were imputed using LOCF approach for subjects who had data for at least one scheduled visit (including Early Termination) subsequent to the baseline measurement. Subjects without post-baseline measurement were categorized as not achieving goal.
Measure: Number; unit: percentage of subjects
Arm/Group | Exenatide Once Weekly | Exenatide Twice Daily
Number analyzed (Participants) | 129 | 123
percentage of subjects | 58.1 | 30.1
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Exenatide Twice Daily; Analysis: Percentages of subjects achieving HbA1c target value of <7% at Week 24 were compared between treatments using a Cochran-Mantel-Haenszel (CMH) test, in which baseline HbA1c stratum (<9% or >=9%) and concomitant SU use at screening served as the stratification factors. Null hypothesis: no difference between treatments in percentage of subjects achieving HbA1c target. Power: based on the primary measurement; Test type: Superiority or Other; p < .0001, Cochran-Mantel-Haenszel — Multiplicity adjustment using Hochberg procedure for the 3 key secondary endpoints (i.e., percent to achieving HbA1c goal of <7%, change in fasting glucose, and percent of achieving fasting plasma glucose goal of <=126 mg/dL) was performed

3. Secondary Outcome: Percentage of Subjects Achieving HbA1c Target of <=6.5%
Description: Percentages of subjects achieving HbA1c target values of <=6.5% at Week 24.
Time Frame: Week 24
Population: as for outcome 2
Measure: Number; unit: percentage of subjects
Arm/Group | Exenatide Once Weekly | Exenatide Twice Daily
Number analyzed (Participants) | 129 | 123
percentage of subjects | 41.1 | 16.3
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Exenatide Twice Daily; Analysis: Percentages of subjects achieving HbA1c target values of <=6.5% at Week 24 were compared between treatments using a CMH test, in which baseline HbA1c stratum (<9% or >=9%) and concomitant SU use at screening served as the stratification factors. Null hypothesis: no difference between treatments in percentage of subjects achieving HbA1c target. Power: based on the primary measurement; Test type: Superiority or Other; p < .0001, Cochran-Mantel-Haenszel

4. Secondary Outcome: Change in Fasting Plasma Glucose From Baseline to Week 24
Description: Change in fasting plasma glucose from baseline (Day 1) to Week 24.
Time Frame: Day 1, Week 24
Population: ITT Population. Missing data up to Week 24 were imputed using LOCF approach for subjects who had data for at least one scheduled visit (including Early Termination) subsequent to the baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Exenatide Once Weekly | Exenatide Twice Daily
Number analyzed (Participants) | 127 | 117
mg/dL | -25.1 (4.32) [-33.6 to -16.6] | -4.6 (4.50) [-13.5 to 4.2]
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Exenatide Twice Daily; Analysis: Change in fasting plasma glucose from baseline (Day 1) to Week 24 was analyzed by an ANCOVA model including treatment, baseline HbA1c stratum (<9% or >=9%), and concomitant SU use at screening as factors, and baseline value of the fasting plasma glucose as a covariate. Null hypothesis: no difference between treatments in change from baseline fasting plasma glucose. Power: based on the primary measurement; Test type: Superiority or Other; p = 0.0006, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -20.4, 95% CI 2-sided [-31.4 to -9.5], Standard Error of Mean 5.57

5. Secondary Outcome: Percentage of Subjects Achieving Fasting Plasma Glucose Target of <=126 mg/dL
Description: Percentages of subjects achieving fasting plasma glucose target of <=126 mg/dL at Week 24.
Time Frame: Week 24
Population: as for outcome 2
Measure: Number; unit: percentage of subjects
Arm/Group | Exenatide Once Weekly | Exenatide Twice Daily
Number analyzed (Participants) | 129 | 123
percentage of subjects | 50.4 | 30.9
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Exenatide Twice Daily; Analysis: Percentages of subjects achieving fasting plasma glucose target of <=126 mg/dL at Week 24 were compared between treatments using a CMH test, in which baseline HbA1c stratum (<9% or >=9%) and concomitant SU use at screening served as the stratification factors. Null hypothesis: no difference between treatments in percentage of subjects achieving fasting plasma glucose target. Power: based on the primary measurement; Test type: Superiority or Other; p = 0.0008, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]

6. Secondary Outcome: Change in Body Weight From Baseline to Week 24
Description: Change in body weight from baseline (Day 1) to Week 24.
Time Frame: Day 1, Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Exenatide Once Weekly | Exenatide Twice Daily
Number analyzed (Participants) | 128 | 120
kg | -2.33 (0.369) [-3.05 to -1.60] | -1.37 (0.386) [-2.13 to -0.61]
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Exenatide Twice Daily; Analysis: Change in body weight from baseline (Day 1) to Week 24 was analyzed by an ANCOVA model including treatment, baseline HbA1c stratum (<9% or >=9%), and concomitant SU use at screening as factors, and baseline value of the body weight as a covariate. Null hypothesis: no difference between treatments in change from baseline body weight. Power: based on the primary measurement; Test type: Superiority or Other; p = 0.0514, ANCOVA; Least Squares Mean Difference = -0.95, 95% CI 2-sided [-1.91 to 0.01], Standard Error of Mean 0.487

7. Secondary Outcome: Change in Sitting Systolic Blood Pressure From Baseline to Week 24
Description: Change in systolic blood pressure from baseline (Day 1) to Week 24.
Time Frame: Day 1, Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Exenatide Once Weekly | Exenatide Twice Daily
Number analyzed (Participants) | 128 | 120
mmHg | -2.9 (1.13) [-5.2 to -0.7] | -1.2 (1.19) [-3.5 to 1.2]
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Exenatide Twice Daily; Analysis: Change in systolic blood pressure from baseline (Day 1) to Week 24 was analyzed by an ANCOVA model including treatment, baseline HbA1c stratum (<9% or >=9%), and concomitant SU use at screening as factors, and baseline value of the systolic blood pressure as a covariate. Null hypothesis: no difference between treatments in change from baseline systolic blood pressure. Power: based on the primary measurement; Test type: Superiority or Other; p = 0.2367, ANCOVA; Least Squares Mean Difference = -1.8, 95% CI 2-sided [-4.7 to 1.2], Standard Error of Mean 1.50

8. Secondary Outcome: Change in Sitting Diastolic Blood Pressure From Baseline to Week 24
Description: Change in diastolic blood pressure from baseline (Day 1) to Week 24.
Time Frame: Day 1, Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Exenatide Once Weekly | Exenatide Twice Daily
Number analyzed (Participants) | 128 | 120
mmHg | 0.2 (0.74) [-1.3 to 1.6] | -0.1 (0.78) [-1.7 to 1.4]
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Exenatide Twice Daily; Analysis: Change in diastolic blood pressure from baseline (Day 1) to Week 24 was analyzed by an ANCOVA model including treatment, baseline HbA1c stratum (<9% or >=9%), and concomitant SU use at screening as factors, and baseline value of the diastolic blood pressure as a covariate. Null hypothesis: no difference between treatments in change from baseline diastolic blood pressure. Power: based on the primary measurement; Test type: Superiority or Other; p = 0.7717, ANCOVA; Least Squares Mean Difference = 0.3, 95% CI 2-sided [-1.7 to 2.2], Standard Error of Mean 0.98

9. Secondary Outcome: Change in Total Cholesterol From Baseline to Week 24
Description: Change in total cholesterol from baseline (Day 1) to Week 24.
Time Frame: Day 1, Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Exenatide Once Weekly | Exenatide Twice Daily
Number analyzed (Participants) | 119 | 104
mg/dL | -15.4 (2.61) [-20.5 to -10.2] | 0.6 (2.79) [-4.9 to 6.1]
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Exenatide Twice Daily; Analysis: Change in total cholesterol from baseline (Day 1) to Week 24 was analyzed by an ANCOVA model including treatment, baseline HbA1c stratum (<9% or >=9%), and concomitant SU use at screening as factors, and baseline value of the total cholesterol as a covariate. Null hypothesis: no difference between treatments in change from baseline total cholesterol. Power: based on the primary measurement; Test type: Superiority or Other; p < .0001, ANCOVA; Least Squares Mean Difference = -16.0, 95% CI 2-sided [-22.9 to -9.1], Standard Error of Mean 3.50

10. Secondary Outcome: Change in High-density Lipoprotein (HDL) From Baseline to Week 24
Description: Change in HDL from baseline (Day 1) to Week 24.
Time Frame: Day 1, Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Exenatide Once Weekly | Exenatide Twice Daily
Number analyzed (Participants) | 119 | 104
mg/dL | 0.0 (0.60) [-1.2 to 1.2] | 1.3 (0.64) [0.0 to 2.5]
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Exenatide Twice Daily; Analysis: Change in HDL from baseline (Day 1) to Week 24 was analyzed by an ANCOVA model including treatment, baseline HbA1c stratum (<9% or >=9%), and concomitant SU use at screening as factors, and baseline value of the HDL as a covariate. Null hypothesis: no difference between treatments in change from baseline HDL. Power: based on the primary measurement; Test type: Superiority or Other; p = 0.1251, ANCOVA; Least Squares Mean Difference = -1.2, 95% CI 2-sided [-2.8 to 0.3], Standard Error of Mean 0.80

11. Secondary Outcome: Ratio of Triglycerides at Week 24 to Baseline
Description: Ratio of triglycerides (measured in mg/dL) at Week 24 to baseline (Day 1). Log (Postbaseline Triglycerides) - log (Baseline Triglycerides); change from baseline to endpoint is presented as ratio of endpoint to baseline.
Time Frame: Day 1, Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Exenatide Once Weekly | Exenatide Twice Daily
Number analyzed (Participants) | 119 | 104
ratio | 0.94 (0.032) [0.88 to 1.00] | 0.99 (0.036) [0.92 to 1.06]
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Exenatide Twice Daily; Analysis: Triglycerides data were logarithm-transformed and the change at Week 30 to baseline (Day 1) , expressed as the ratio, was analyzed by an ANCOVA model including treatment, baseline HbA1c stratum (<9% or >=9%), and concomitant SU use at screening as factors, and baseline value of the triglycerides as a covariate. Null hypothesis: no difference between treatments in change from baseline triglycerides. Power: based on the primary measurement; Test type: Superiority or Other; p = 0.2558, ANCOVA; Geometric Least Squares Mean Ratio = 0.95, 95% CI 2-sided [0.87 to 1.04], Standard Error of Mean 0.043

12. Secondary Outcome: Assessment on Event Rate of Treatment-emergent Major Hypoglycemic Events
Description: The major hypoglycemia category included events that, in the judgment of the investigator or physician, resulted in loss of consciousness, seizure, coma, or other change in mental status consistent with neuroglycopenia, in which symptoms resolved after administration of intramuscular glucagon or intravenous glucose, required third-party assistance, and was accompanied by a blood glucose concentration of less than 54 mg/dL prior to treatment, whether or not symptoms of hypoglycemia were perceived by the subject.
Time Frame: Day 1 to Week 24
Population: ITT Population. Analysis was done for SU ITT patients (ITT patients taking SU) and Non-SU ITT patients separately.
Measure: Mean (Standard Error); unit: rate per subject-year
Groups:
- Exenatide Once Weekly With SU: Subjects with subcutaneous injection of 2 mg exenatide, once a week using concomitant SU at screening
- Exenatide Twice Daily With SU: Subjects with subcutaneous injection of exenatide, twice a day (5 mcg exenatide per dose for first 4 weeks, then 10 mcg exenatide per dose for 20 weeks) using concomitant SU at screening
- Exenatide Once Weekly No SU: Subjects with subcutaneous injection of 2 mg exenatide, once a week not using concomitant SU at screening
- Exenatide Twice Daily No SU: Subjects with subcutaneous injection of exenatide, twice a day (5 mcg exenatide per dose for first 4 weeks, then 10 mcg exenatide per dose for 20 weeks) not using concomitant SU at screening
Arm/Group | Exenatide Once Weekly With SU | Exenatide Twice Daily With SU | Exenatide Once Weekly No SU | Exenatide Twice Daily No SU
Number analyzed (Participants) | 40 | 34 | 89 | 89
rate per subject-year | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000)

13. Secondary Outcome: Assessment on Event Rate of Treatment-emergent Minor Hypoglycemic Events
Description: The minor hypoglycemia category included events in which symptoms consistent with hypoglycemia were accompanied by a blood glucose concentration of less than 54 mg/dL prior to treatment and not classified as major hypoglycemia.
Time Frame: Day 1 to Week 24
Population: ITT Population. Analysis was done for SU ITT patients (ITT patients taking SU) and Non-SU ITT patients separately.
Measure: Mean (Standard Error); unit: rate per subject-year
Arm/Group | Exenatide Once Weekly With SU | Exenatide Twice Daily With SU | Exenatide Once Weekly No SU | Exenatide Twice Daily No SU
Number analyzed (Participants) | 40 | 34 | 89 | 89
rate per subject-year | 0.75 (0.217) | 0.31 (0.153) | 0.00 (0.000) | 0.00 (0.000)

ADVERSE EVENTS:
Arm/Group | Exenatide Once Weekly | Exenatide Twice Daily
Serious Adverse Events (participants affected / at risk) | 3/129 | 5/123
Other Adverse Events (participants affected / at risk) | 44/129 | 58/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide Once Weekly (N=129) | Exenatide Twice Daily (N=123)
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide Once Weekly (N=129) | Exenatide Twice Daily (N=123)
Nausea (Gastrointestinal disorders) | 18 | 43
Diarrhoea (Gastrointestinal disorders) | 12 | 5
Upper respiratory tract infection (Infections and infestations) | 9 | 5
Injection site erythema (General disorders) | 7 | 3
Headache (Nervous system disorders) | 6 | 10
Vomiting (Gastrointestinal disorders) | 6 | 11
Dizziness (Nervous system disorders) | 3 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less